CLINICAL TRIAL: NCT05527769
Title: Prospective Study Evaluating Postoperative Pain and Functional Recovery After Mastectomy and Immediate Breast Reconstruction by Implant: Prepectoral Versus Subpectoral Technique
Brief Title: Pain and Functional Recovery After Mastectomy and IBR by Implant: Prepectoral Versus Subpectoral Technique
Acronym: DREAM-RMI
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2021-36
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-pectoral prosthesis: breast cancer patients with an indication for total mastectomy + immediate breast reconstruction (IBR) by prosthesis using a pre-pectoral technique
  Interventions: Procedure: mastectomy + immediate breast reconstruction
- retropectoral prosthesis: breast cancer patients with an indication for total mastectomy + immediate breast reconstruction (IBR) by prosthesis using the retropectoral technique
  Interventions: Procedure: mastectomy + immediate breast reconstruction

INTERVENTIONS:
Procedure: mastectomy + immediate breast reconstruction — pre- or retro pectoral prosthesis

SUMMARY:
This is a prospective, single-center, non-randomized study of immediate breast reconstruction (IBR) using a pre- or retro-pectoral technique in patients with breast cancer who have undergone total mastectomy.

The technique used is chosen according to the characteristics of the breast, the morphology of the patient and her wishes after informed information on the different techniques. The aim is not to compare the two techniques but rather to evaluate the early functional results of these two methods in order to better understand them and to propose a management adapted to each.

The main objective will be to evaluate the postoperative pain by BPI questionnaire.

The investigators also wish to observe the functional results of the homolateral upper limb by DASH questionnaire, the quality of life by BREAST Q questionnaire and the occurrence of complications.

DETAILED DESCRIPTION:
describe the occurrence of complications between pre-pectoral and retro-pectoral technique in patients with breast cancer who have total mastectomy.

evaluate the postoperative pain by Brief Pain Inventory (BPI) self assesment observe the functional results of the homolateral upper limb by Disabilities of the Arm, Shoulder and Hand (DASH) self assesment observe quality of life by BREAST Q questionary

ELIGIBILITY:
Inclusion Criteria:

1. Major patients
2. With breast cancer and indication for total mastectomy
3. With a desire for immediate breast reconstruction
4. Total mastectomy procedure and Immediate Breast Reconstruction by Pre-pectoral or Retro-Pectoral prosthesis
5. Information of the patient and collection of his/her non-opposition
6. Affiliation with a social securitý scheme, or beneficiary of such a scheme

Exclusion Criteria:

1. Prophylactic mastectomies
2. Metastatic patients
3. Patients requiring another surgical technique
4. Person in an emergency situation, person of legal age under legal protection (adult under guardianship, curators or safeguard of justice), or unable to express consent,
5. Impossibility to submit to the medical follow-up of the trial for geographical, social or psychological reasons
6. Pregnant or likely to be pregnant

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Major patients followed for breast cancer with indication of mastectomy with immediate breast reconstruction by prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Describe postoperative pain and functional results | 6 month
  Brief Pain Inventory (BPI) short form - 4 scales from 1 (No pain) to 10 (max pain) + 7 scales from 1 (no discomfort) to 10 (max discomfort) to determine if the pain interfered with activities of daily living

SECONDARY OUTCOMES:
Assessing quality of life and aesthetic satisfaction | 6 months
  breast questionary pre-post operative reconstruction module
Evaluate the function of the homolateral upper limb | 6 months
  Disabilities of the Arm, Shoulder and Hand self-assessment
Describe the occurrence of postoperative complications | 3 months
  postoperative complications
Describe the length of operative stay (for the initial reconstruction), for all patients and according to the methods of reconstruction performed | 3 months
  duration of hospitalization
Describe the duration of drainage for all patients and according to the methods of reconstruction performed | 3 months
  duration of drainage in the breast and back, number of punctures and total volume of seroma punctures (classification <2)
Describe the number of surgery(s) required to obtain a good aesthetic result | 3 months
  number of surgery(s)
Describe the number of consultations for seroma punctures, for all patients and according to the methods of reconstruction performed | 3 months
  number of punctures and total volume of seroma punctures (classification <2)

CONTACTS AND LOCATIONS:
Overall Officials: Céline RENAUDEAU, MD, Principal Investigator — celine.renaudeau@ico.unicancer.fr
Locations (1):
- Institut de Cancerologie de L'Ouest, Saint-Herblain, France